CLINICAL TRIAL: NCT00302900
Title: Preventing Adverse Reactions in Novice Blood Donors
Brief Title: Preventing Negative Reactions in First Time Blood Donors to Encourage Subsequent Blood Donations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 371; R01HL077438 (NIH)
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2009-02

CONDITIONS: Syncope, Vasovagal
Keywords: Blood Donation; Syncope; Vasovagal Reactions
MeSH Terms: conditions — Syncope, Vasovagal; Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Pre-donation water and muscle tension during donation
  Interventions: Behavioral: Pre-Donation Water Consumption; Behavioral: Muscle Tensing Exercise During Donation
- 2 (Experimental): Pre-donation water
  Interventions: Behavioral: Pre-Donation Water Consumption
- 3 (Sham Comparator): Pre-donation muscle tension
  Interventions: Behavioral: Muscle Tensing Exercise Prior to Donation
- 4 (No Intervention): Standard donation

INTERVENTIONS:
Behavioral: Pre-Donation Water Consumption — Consumption of 500 ml of bottled water 30 minutes prior to donating
  Arms: 1; 2
Behavioral: Muscle Tensing Exercise During Donation — Alternating leg lifts at 10-second intervals during donation
  Arms: 1
Behavioral: Muscle Tensing Exercise Prior to Donation — Alternating leg lifts at 10-second intervals prior to insertion of the donation needle
  Arms: 3

SUMMARY:
Many individuals experience negative reactions when donating blood, including dizziness, lightheadedness, or fainting. Such reactions may discourage them from donating again. This study will evaluate the effectiveness of pre-donation water consumption and a muscle tensing exercise during donation to reduce negative reactions among new blood donors. This study will also evaluate whether reducing negative reactions increases the likelihood of donors returning to give blood in the future.

DETAILED DESCRIPTION:
Severe and potentially dangerous shortages in the blood supply are increasingly common in the United States. As the population ages and as more stringent donor eligibility restrictions are enforced, blood shortages are expected to worsen. One way to meet the increasing demand for blood is to recruit new blood donors. Ideally, these individuals would become lifelong donors, and contribute up to six times per year and up to hundreds of units of blood within a lifetime. Unfortunately, less than half of all new donors provide a second donation. Many individuals who donate blood experience dizziness, weakness, lightheadedness, or in severe cases, fainting. As a result of these negative reactions, many individuals never donate blood again. Preventing these reactions may be an effective way to encourage subsequent blood donations. The purpose of this study is to evaluate the effectiveness of consuming water prior to donation and performing a muscle tensing exercise during donation as ways to reduce negative reactions in new blood donors. The study's long-term goal is to provide blood collection agencies with simple and inexpensive strategies to prevent negative reactions and enhance donor retention.

This study will enroll American Red Cross blood donors who have donated blood no more than twice previously. Participants will be randomly assigned to one of the following four groups: 1) pre-donation water consumption and muscle tensing exercise during donation; 2) pre-donation water consumption; 3) pre-donation muscle tensing exercise; or 4) no treatment. Participant reactions will be assessed at the time of donation by self-report and phlebotomist ratings, as well as by self-report 24 hours following the donation. Participants' subsequent donation history will be tracked for two years by reviewing the American Red Cross national donor database.

ELIGIBILITY:
Inclusion Criteria:

* Must meet American Red Cross donor eligibility requirements

Exclusion Criteria:

* No more than two prior blood donations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2006-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Participant ratings of negative (vasovagal) reactions | Measured within 30 minutes of donating
Phlebotomist ratings of donor reactions | Measured immediately following donation
Number of repeat donations | Measured 2 years post-donation

SECONDARY OUTCOMES:
Subjective ratings of muscle soreness and fatigue | Measured 24 hours post-donation
Negative (vasovagal) reactions | Measured 24 hours post-donation

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. France, PhD, Principal Investigator — Ohio University
Locations (2):
- United States (2):
  - Ohio University, Athens, Ohio
  - American Red Cross Blood Services - Central Ohio Region, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data is available upon request from the primary investigator.